CLINICAL TRIAL: NCT00019396
Title: Phase II Study of Flt3 Ligand Alone or in Combination With Melanoma Peptide Immunization in Patients With Metastatic Melanoma or Renal Cell Cancer
Brief Title: flt3L With or Without Vaccine Therapy in Treating Patients With Metastatic Melanoma or Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065997; NCI-98-C-0040; NCI-T97-0092; NCT00001687 (obsolete NCT alias)
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Stage IV Melanoma; Stage IV Renal Cell Cancer; Recurrent Renal Cell Cancer; Recurrent Melanoma
Keywords: adult solid tumor; body system/site cancer; cancer; kidney tumor; kidney/urinary cancer; melanoma; recurrent melanoma; recurrent renal cell cancer; renal cell cancer; skin tumor; solid tumor; stage IV melanoma; stage IV renal cell cancer; stage, melanoma; stage, renal cell cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Neoplasms; Urologic Neoplasms; Skin Neoplasms | interventions — flt3 ligand protein; MART-1 Antigen; montanide ISA 51

INTERVENTIONS:
Drug: flt3 ligand
Drug: gp100 antigen
Drug: MART-1 antigen
Drug: Montanide ISA-51
Drug: tyrosinase peptide

SUMMARY:
RATIONALE: The drug flt3L may stimulate a person's immune system and help to kill tumor cells. Vaccines made from melanoma cells may make the body build an immune response to and kill their tumor cells.

PURPOSE: Phase II trial to study the effectiveness of flt3L with or without vaccine therapy in treating patients with metastatic melanoma or renal cell cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the immunologic and biologic activity of flt3 ligand (Flt3L) alone in patients with metastatic renal cell cancer or HLA-A2.1 negative melanoma.

II. Evaluate the immunologic and biologic activity of Flt3L alone or in combination with melanoma peptide immunization (MART-1, gp100:209-217, gp100:280-288, and tyrosinase) in patients with metastatic, HLA-A2.1 positive melanoma.

PROTOCOL OUTLINE: Patients are assigned to 1 of 3 treatment groups:

Group 1 (renal cell cancer): Patients receive Flt3 ligand (Flt3L) subcutaneously (SQ) alone on days 1-14.

Group 2 (HLA-A2.1 negative melanoma): Patients receive Flt3L SQ alone on days 1-14.

Group 3 (HLA-A2.1 positive melanoma): Patients may receive either Flt3L SQ alone on days 1-14 or in combination with melanoma peptide immunization. Patients may receive melanoma peptide immunization comprised of MART-1 immunodominant peptide, gp100:209-217, gp100:280-288, and tyrosinase peptide emulsified in Montanide ISA-51 SQ on day 12 of Flt3L administration.

Treatment repeats every 4 weeks for 2 courses. Patients with no response or minor response may receive 2 additional courses. Patients with disease progression after 1 course are removed from study.

PROJECTED ACCRUAL:

Approximately 54-96 patients (18-32 per treatment group) will be accrued for this study within 16 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically proven metastatic melanoma or renal cell cancer Patients receiving melanoma peptide immunizations must be HLA-A2.1 positive Measurable disease --Prior/Concurrent Therapy-- Biologic therapy: At least 1 month since prior biologic therapy Chemotherapy: At least 1 month since prior chemotherapy Endocrine therapy: No concurrent systemic steroid therapy At least 1 month since prior steroid therapy Radiotherapy: At least 1 month since prior radiotherapy Surgery: Prior surgery allowed Other: Greater than 1 month since prior therapy --Patient Characteristics-- Age: Not specified Performance Status: ECOG 0-1 Life Expectancy: Greater than 3 months Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 90,000/mm3 No coagulation disorders Hepatic: Bilirubin no greater than 1.6 mg/dL AST and ALT less than 2 times normal Renal: Creatinine no greater than 2 mg/dL Cardiovascular: No major cardiovascular disease Pulmonary: No major pulmonary disease Other: Not pregnant or nursing Negative pregnancy test HIV negative Hepatitis B surface antigen negative No allergic reaction to Montanide ISA-51 No active systemic infection No prior autoimmune disorders

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-02; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Hwu, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States